CLINICAL TRIAL: NCT07059104
Title: Implant-based Breast Surgery and Reconstruction Following Bariatric Surgery: an Observational Register-based Study on Prevalence and Risk Factors for Surgical Complications
Brief Title: Implant-based Breast Reconstruction in Post-bariatric Women - a Registry-based National Study
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 284398
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Reconstruction; Bariatric Surgery; Breast Implant; Breast Implant Infection; Surgical Complication; Mastopexy; Weight Loss
Keywords: plastic surgery; breast augmentation; breast implant; augmentation mastopexy; complications; post-bariatric reconstruction
MeSH Terms: conditions — Breast Neoplasms; Weight Loss | interventions — Breast Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breast implant after weight loss surgery: Women who have had weight loss surgery and are having breast plastic surgery (benign)
  Interventions: Procedure: Breast augmentation
- Breast implant controls: Women who have not had weight loss surgery and are having breast plastic surgery (benign)
  Interventions: Procedure: Breast augmentation
- Breast reconstruction after weight loss surgery: Women who have had weight loss surgery and are having breast reconstruction after mastectomy (malignant)
  Subgroups: therapeutic mastectomies, risk-reducing mastectomies,immediate breast reconstruction, delayed breast reconstruction.
  Interventions: Procedure: Breast reconstruction after mastectomy
- Breast reconstruction controls: Women who have not had weight loss surgery and are having breast reconstruction after mastectomy (malignant).Subgroups: therapeutic mastectomies, risk-reducing mastectomies, immediate breast reconstruction, delayed breast reconstruction.
  Interventions: Procedure: Breast reconstruction after mastectomy

INTERVENTIONS:
Procedure: Breast augmentation — Breast augmentation with an implant
  Other Names: Breast enlargement; Augmentation mastopexy; breast implant; post-bariatric breast reconstruction
  Groups: Breast implant after weight loss surgery; Breast implant controls
Procedure: Breast reconstruction after mastectomy — Breast reconstruction after mastectomy
  Other Names: DIEP flap; implant-based breast reconstruction; risk reducing mastectomy; immediate breast reconstruction; delayed breast reconstruction; autologous breast reconstruction; therapeutic mastectomy
  Groups: Breast reconstruction after weight loss surgery; Breast reconstruction controls

SUMMARY:
The goal of this national registry-based study is to investigate the prevalence of reconstructive breast surgery and risk factors for surgical complications in women who have had weight loss surgery previously. The main questions it aims to answer are:

1. What is the perceived need for breast implants after weight loss surgery, described as the proportion who have breast implants, and what characteristics, in terms of demographics and surgical details, do the operated women have?
2. In women who have breast enlargement or breast enlargement combined with a lift, are there any differences between the women who have had weight loss surgery and other women regarding complications after the operation and characteristics of the surgery, for example skin incision and choice of implant (for example texture, shape, size)?
3. In women who have delayed breast reconstruction after breast cancer, that is have had their breast/s reconstructed in a separate operation, are there any differences between the women who have had weight loss surgery and other women regarding complications after the operation and characteristics of the surgery, for example in technique used (autologous versus implant-based, choice of implant, such as texture, shape and size), and timing of the surgery? Immediate breast reconstruction is defined as performed at the same time as the mastectomy, and delayed as an operation performed later in a separate operation.
4. In women who have immediate breast reconstruction after breast cancer?, that is have a breast reconstruction at the same time as the mastectomy, are there any differences between the women who have had weight loss surgery and other women regarding complications after the operation and characteristics of the surgery, for example in technique used (autologous versus implant-based, choice of implant, such as texture, shape and size), and timing of the surgery? Immediate breast reconstruction is defined as performed at the same time as the mastectomy, and delayed as an operation performed later in a separate operation.
5. In women who have risk reducing mastectomies, are there any differences between he women who have had weight loss surgery and other women regarding complications after the operation and characteristics of the surgery, for example in technique used (autologous versus implant-based, choice of implant, such as texture, shape and size), and timing of the surgery? Immediate breast reconstruction is defined as performed at the same time as the mastectomy, and delayed as an operation performed later in a separate operation.
6. Are there any identifiable risk factors for complications after breast reconstructive surgery, specific to the women who have had weight loss surgery and other women?

Researchers will compare the patients to women who have the same type of reconstructive breast surgery but have not had bariatric surgery previously.

The study will use prospectively collected data from seven registers: The Scandinavian Obesity Surgery Register (SOReg), The Swedish Breast Implant Register (BRIMP), the Swedish National Quality Register for Breast Cancer (NKBC), the Swedish National Diabetes Register (NDR), Statistics Sweden (SCB), the Swedish inpatient register, and the Swedish National Prescribed Drug Register.

ELIGIBILITY:
Inclusion Criteria:

Inclusion in Soreg and thereafter inclusion in either BRIMP or NKBC

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who have weight loss surgery and then have breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of breast plastic surgery following bariatric surgery | 10 years. The time frame is longer than the study duration, as it is based on already collected registry-based data.
  How many of the women who have bariatric surgery later have breast plastic surgery according to national registries.
Demography | 3 months
  Demography of the patients compared to the controls (eg. age, BMI, education level, income level, marital status, country of origin, county of residence, employment status, co-morbidity, usage of drugs)
Surgical details | 3 months
  All surgical details given in BRIMP and in NKBC, eg type of implant, type of reconstruction etc.
Complications and risk factors for complications | 10 years
  Complications following the surgery and risk factors as defined in the national registers.
Re-operations and risk factors for re-operations | 10 years
  Any re-operations and risk factors registered in the national registries.

SECONDARY OUTCOMES:
Drugs | 6 months
  Usage of anticoagulants, pain killers, and antibiotics 3 months before and 3 months after the breast operation.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hansson, professor, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Västra Götalandsregionen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansson E, Li Y, Grimby-Ekman A, Elander A, Paganini A. Nomogram Risk Prediction Model for Reoperation/Revision in the First 5 Years After Primary Breast Augmentation Following Massive Weight Loss: A Clinical Tool. Aesthet Surg J. 2025 Nov 11:sjaf234. doi: 10.1093/asj/sjaf234. Online ahead of print. PMID 41219167
- [Derived] Paganini A, Ottosson J, Halle M, Mirzaei N, Gudbjornsdottir S, Grimby-Ekman A, Hansson E. Frequency, demographics, and comorbidity of women with post-bariatric breast implants: A Swedish population-based controlled study. J Plast Reconstr Aesthet Surg. 2025 Dec;111:145-155. doi: 10.1016/j.bjps.2025.10.004. Epub 2025 Oct 8. PMID 41151312